CLINICAL TRIAL: NCT06011616
Title: Effects of Upperlimb Sensorimotor Training in Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/Letter-014194
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 2 group parallel randomized control trial; both groups will be recruited and provided with interventions in parallel
Who Masked: Participant
Masking Description: Only the subjects would be masked about the group they belong too.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): Superficial and Deep Sensory training: 5 sets of 9 min, 3 times a week for 8 weeks.
  Motor training: 5 sets of 9 min, 3 times a week for 8 weeks. Conventional therapy: 30 min, 3 days for 8 weeks
  Interventions: Other: Sensory training; Other: Motor training; Other: Conventional exercises
- control group (Active Comparator): Motor training: 5 sets of 9 min, 3 times a week for 8 weeks. Conventional therapy: 30 min, 3 days for 8 weeks
  Interventions: Other: Motor training; Other: Conventional exercises

INTERVENTIONS:
Other: Sensory training — sensory training includes superficial sensory and deep sensory activities i.e. play with dough, painting with finger, recognizing objects with blocked vision, recognizing the drawn figure on palm, oint compression, bearing the weight on the paretic hand, leaning on the paretic side, walking with hand, rolling the heavy objects, dough squeezing etc.
  Arms: interventional group
Other: Motor training — Motor training would involve activitoes such as throwing and catching a ball, targeted ball throwing, hand in hand ball transferring, ball rolling, hitting a ball to ground and wall, hand roller etc.
Other: Conventional exercises — stretching exercises, muscle strengthening exercises, static weight bearing exercises, positioning

SUMMARY:
The study aims to determine the effects of upper limb sensorimotor training as compared to task oriented raining in subjects with cerebral palsy. The study will target the upperlimb functions using multiple outcomes and will find the changes in subjects undergoing sensorimotor or task oriented training.

DETAILED DESCRIPTION:
The stduy will include subjects fulfilling the inclusion criteria, will be divided into 2 groups; interventional and control. The interventional group will be recieving sensorimotor training comprising of sensory activities and motor activities. The control group will be having motor activities in the form of task oriented training. The duration of intervention would be 40 minutes in each group, 3 days a week, for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic cerebral palsy Modified Ashworth scale score 2 and 3

Exclusion Criteria:

* Other neurological disorders Previous upper limb surgeries Botox injection in last 1 year

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline
  Modified Ashworth Scale measures the level of spasticity, ranging from 0-4 with 0 being no increase in tone and 4 being affected parts rigid in flexion
Modified Ashworth Scale (MAS) | After 4 weeks
  Modified Ashworth Scale measures the level of spasticity, ranging from 0-4 with 0 being no increase in tone and 4 being affected parts rigid in flexion
Modified Ashworth Scale (MAS) | After 8 weeks
  Modified Ashworth Scale measures the level of spasticity, ranging from 0-4 with 0 being no increase in tone and 4 being affected parts rigid in flexion
Finger Joint Position Sense | Baseline
  Finger Joint Position Sense is done to determine the sense of position, in whcih the subjet's finger is moved by the outcome assesser with eyes closed.
Finger Joint Position Sense | After 4 weeks
  Finger Joint Position Sense is done to determine the sense of position, in whcih the subjet's finger is moved by the outcome assesser with eyes closed.
Finger Joint Position Sense | After 8 weeks
  Finger Joint Position Sense is done to determine the sense of position, in whcih the subjet's finger is moved by the outcome assesser with eyes closed.
Manual ability classification system | Baseline
  Manual ability classification system is used to determine daily use hand activities
Manual ability classification system | After 4 weeks
  Manual ability classification system is used to determine daily use hand activities
Manual ability classification system | After 8 weeks
  Manual ability classification system is used to determine daily use hand activities
Manual Muscle Testing | Baseline
  Manual Muscle Testing is used to determine the strength. the score varies from 0-5; 0 means no contraction and 5 means movement aagainst maximum resistance
Manual Muscle Testing | After 4 weeks
  Manual Muscle Testing is used to determine the strength. the score varies from 0-5; 0 means no contraction and 5 means movement aagainst maximum resistance
Manual Muscle Testing | After 8 weeks
  Manual Muscle Testing is used to determine the strength. the score varies from 0-5; 0 means no contraction and 5 means movement aagainst maximum resistance
Abilities of Hand (ABILHAND-KIDS) | Baseline
  This tool is used to determine the hand and manual abilities of the kids. It has 21 manual activites with 3 levels each; 1 as impossible, 2 difficult and 3 easy.
Abilities of Hand (ABILHAND-KIDS) | After 4 weeks
  This tool is used to determine the hand and manual abilities of the kids. It has 21 manual activites with 3 levels each; 1 as impossible, 2 difficult and 3 easy.
Abilities of Hand (ABILHAND-KIDS) | After 8 weeks
  This tool is used to determine the hand and manual abilities of the kids. It has 21 manual activites with 3 levels each; 1 as impossible, 2 difficult and 3 easy.
Pediatric Arm Function Test | Baseline
  This is used to determine the upper extremity movement patterns in playful situation. It has 26 items with each at 6 levels ranging from minimum to maximum function.
Pediatric Arm Function Test | After 4 weeks
  This is used to determine the upper extremity movement patterns in playful situation. It has 26 items with each at 6 levels ranging from minimum to maximum function.
Pediatric Arm Function Test | After 8 weeks
  This is used to determine the upper extremity movement patterns in playful situation. It has 26 items with each at 6 levels ranging from minimum to maximum function.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khushnood, MSNMPT, Study Chair — Riphah International University
Locations (1):
- Alfarabi Special Education Centre/ Physical Health Centre, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No